CLINICAL TRIAL: NCT00778622
Title: The Relationship Between Baseline Body Weight and Glycemic Control Following Metformin Extended-Release Tablets (Glucophage XR) Monotherapy in Chinese Patients With Newly Diagnosed Type 2 Diabetes
Brief Title: Body Weight Effects on Glucophage's Efficacy in Chinese Diagnosed T2DM Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV138-097
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Results first posted 2013-08-20 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A1 (Experimental): Normal Weight by Body Weight Index
  Interventions: Drug: Metformin XR
- A2 (Experimental): Overweight by Body Weight Index
  Interventions: Drug: Metformin XR
- A3 (Experimental): Obese by Body Weight Index
  Interventions: Drug: Metformin XR

INTERVENTIONS:
Drug: Metformin XR — Tablets, Oral, 500mg tid, 1500 mg/day, 16 weeks

SUMMARY:
The purpose of this study is to investigate the effect of the baseline body mass index (BMI) on the response to Glucophage XR monotherapy in glycemic control in Chinese patients with newly diagnosed type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Age≥ 17 and <80 years,
* Newly diagnosed T2DM (defined as T2DM diagnosed within 6 months prior to enrollment)
* Oral antidiabetic agents naïve (defined as without receiving any anti-diabetic medication therapy before, or having received anti-diabetic medication ≤ 14 days but not received any antidiabetic medication within the last 1 month prior to enrollment)
* HbA1c ≥ 7.0% and ≤10.0%

Exclusion Criteria:

* Women of child bearing potential
* body mass index (BMI)≥35 Kg/m2 or BMI <18.5 Kg/m2
* Hemoglobin A1c (HbA1c)>10.0% or <7.0%
* Active liver disease and/or significant abnormal liver function
* Acute or chronic metabolic acidosis, including diabetic ketoacidosis, with or without coma
* Congestive heart failure defined as New York Heart Association (NYHA) class III or IV and /or left ventricular ejection fraction ≤40%
* Significant cardiovascular history with the past 6 months
* Severe retinopathy, persistent uncontrolled hypertension (SBP≥180mmHg, or DBP≥105mmHg)
* Severe chronic gastrointestinal disease
* History of alcohol abuse or illegal drug abuse within the past 12 months
* Diagnosed anemia
* Creatine kinase ≥3 X ULN
* Serum creatinine ≥1.5 mg/dL(133μmol/L) [males], ≥1.4 mg/dL(124 μmol/L)[females]
* Alanine amino transferase (ALT) and/or aspartate amino transferase (AST)> 1.5 X ULN and/or total bilirubin > 2 X ULN
* Hemoglobin <12g/dL [males], <11g/dL [females]
* Allergies and Adverse Drug Reactions
* Prohibited Treatments and/or Therapies
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness
* Subjects decline to participate

Ages: 17 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- China (4):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangdong Province, Guangdong
  - Local Institution, Guangdong, Guangdong
  - Local Institution, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Ji L, Li H, Guo X, Li Y, Hu R, Zhu Z. Impact of baseline BMI on glycemic control and weight change with metformin monotherapy in Chinese type 2 diabetes patients: phase IV open-label trial. PLoS One. 2013;8(2):e57222. doi: 10.1371/journal.pone.0057222. Epub 2013 Feb 28. PMID 23468941
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Started November 2009, Completed March 2011 at Peking University People's Hospital. Participants diagnosed with Type 2 diabetes mellitus 6 months prior to enrollment; were oral antidiabetic agent naive (either having received no antidiabetic agents or received agents 14 days or less, or received none within a month of enrollment in the study.
Pre-assignment Details: Participants had glycosated hemoglobin A1c (HbA1c) screening values greater than, equal to 7.0% and less than, equal to 10.0%. Participants were between the ages of 17 and 80 years of age and Chinese Asian. Screening visit was up to 7 days prior to Day 1 (treatment).
Groups:
- Glucophage XR in Normal Weight Participants: Normal weight was defined as body mass index (BMI) greater than, equal to (>=)18.5 kilogram per meter squared (kg/m^2) and less than (<) 24 kg/m^2. Initial dose of Glucophage extended release (XR) on Day 1 was 500 mg taken once daily orally with the evening meal. Drug was titrated up by increments of 500 mg each week to a maximum dose of 2000 mg at Week 4 and for the remaining treatment if the fasting plasma glucose (FPG) was greater than 7.0 mmol/L (126 mg/dL). If the FPG was more than 10.0 mmol/L (greater than 180 mg/dL) at Weeks 4, 8, or 12 and the values were confirmed at a repeated measurement, the participant was discontinued from the treatment. Participants were dosed for a total of 16 weeks.
- Glucophage XR in Overweight Participants: Overweight was defined as body mass index (BMI) greater than, equal to (>=) 24 kg/m^2 and less than (<) 28 kg/m^2. Initial dose of Glucophage extended release (XR) on Day 1 was 500 mg taken once daily orally with the evening meal. Drug was titrated up by increments of 500 mg each week to a maximum dose of 2000 mg at Week 4 and for the remaining treatment if the fasting plasma glucose (FPG) was greater than 7.0 mmol/L (126 mg/dL). If the FPG was more than 10.0 mmol/L (greater than 180 mg/dL) at Weeks 4, 8, or 12 and the values were confirmed at a repeated measurement, the participant was discontinued from the treatment. Participants were dosed for a total of 16 weeks
- Glucophage XR in Obese Participants: Obese was defined as body mass index (BMI) greater than, equal to (>=) 28 kg/m^2. Initial dose of Glucophage extended release (XR)on Day 1 was 500 mg taken once daily orally with the evening meal. Drug was titrated up by increments of 500 mg each week to a maximum dose of 2000 mg at Week 4 and for the remaining treatment if the fasting plasma glucose (FPG) was greater than 7.0 mmol/L (126 mg/dL). If the FPG was more than 10.0 mmol/L (greater than 180 mg/dL) at Weeks 4, 8, or 12 and the values were confirmed at a repeated measurement, the participant was discontinued from the treatment. Participants were dosed for a total of 16 weeks
Period: Overall Study
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Started | 125 | 122 | 124
Completed | 109 | 107 | 109
Not Completed | 16 | 15 | 15
Not completed — Adverse Event | 5 | 4 | 7
Not completed — Withdrawal by Subject | 4 | 5 | 5
Not completed — Lost to Follow-up | 3 | 3 | 2
Not completed — Protocol Violation | 0 | 3 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — immigration | 1 | 0 | 0
Not completed — Other | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population consisted of: all participants enrolled into one of three body weight arms, normal, overweight or obese, based on body mass index at screening; and who were assigned to treatment with Glucophage XR. This population was used for analysis of demographics.
Groups:
- Glucophage XR in Normal Weight Participants: Normal weight was defined as body mass index (BMI) greater than, equal to 18.5 kg/m^2 and < 24 kg/m^2 ). Glucophage XR titrated from Day 1 to Week 4 in increments of 500 mg up to maximum dose of 2000 mg. Participants were dosed for a total of 16 weeks.
- Glucophage XR in Overweight Participants: Overweight was defined as body mass index (BMI) greater than, equal to 24 kg/m^2 and less than 28 kg/m^2. Glucophage XR titrated from Day 1 to Week 4 in increments of 500 mg up to maximum dose of 2000 mg. Participants were dosed for a total of 16 weeks.
- Glucophage XR in Obese Participants: Obese was defined as body mass index (BMI) greater than, equal to 28 kg/m^2. Glucophage XR titrated from Day 1 to Week 4 in increments of 500 mg up to maximum dose of 2000 mg. Participants were dosed for a total of 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants | Total
Number analyzed (Participants) | 125 | 122 | 124 | 371
Age Continuous [Median (Full Range); unit: years] | 53.0 (10.32) [28 to 77] | 51.0 (9.21) [32 to 77] | 52.5 (10.97) [23 to 74] | 52.0 (10.17) [23 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 45 | 52 | 161
  Male | 61 | 77 | 72 | 210
Region of Enrollment [Number; unit: participants]
  China | 125 | 122 | 124 | 371

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline at Week 16 (95% Confidence Interval) in Glycosated Hemoglobin A1c (HbA1c) (Last Observation Carried Forward) - Full Analysis Set (FAS)
Description: Baseline for HbA1c is defined as that value obtained at screening visit. HbA1c was measured as a percent (%) of hemoglobin; normal range was 4.7 to 6.4% and values were obtained through a central laboratory. The Last Observation Carried Forward (LOCF) data set includes data recorded at a given visit or, if no observation is recorded at that visit, data carried forward from the previous visit.
Time Frame: Baseline to Week 16
Population: Full Analysis Set included participants who were enrolled, took at least 1 study medication and had at least 1 post baseline HbA1c assessment. Baseline data was not carried forward or averaged with on-treatment data to impute missing values for the LOCF data set.
Measure: Mean (95% Confidence Interval); unit: percentage of hemoglobin
Groups:
- Glucophage XR in Normal Weight Participants: Normal weight defined as BMI >= 18.5 kg/m^2 and < 24 kg/m^2 .
- Glucophage XR in Overweight Participants: Overweight defined as BMI >= 24 kg/m^2 and < 28 kg/m^2.
- Glucophage XR in Obese Participants: Obese was defined as BMI >= 28 kg/m^2.
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 111 | 111 | 112
percentage of hemoglobin | -1.95 (0.922) [-2.12 to -1.77] | -1.79 (0.941) [-1.96 to -1.61] | -1.68 (0.854) [-1.83 to -1.52]
Statistical Analysis 1: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants vs Glucophage XR in Obese Participants; Standard deviation assumed for changes from baseline in HbA1c maximally was 1.0 across the baseline BMI subgroups. 97 participants in a single subgroup would be sufficient to estimate mean change in HbA1c with precision of 0.20% within the subgroup. Given number of baseline BMI subgroups and no correction for reason of multiplicity was made to the 95% CI within each BMI subgroup, total sample size calculated as 291. Sample size used the method "CI for mean for one group" in nQuery Advisor v6.0; Test type: Superiority or Other; p = 0.0806, ANCOVA — Interpretation based on 2-sided 5% significance level; Change from baseline in HbA1c at Week 16 was dependent variable, BMI was fixed main effect, baseline HbA1c was covariate
Statistical Analysis 2: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants; Test type: Superiority or Other; p = 0.1984, t-test, 2 sided — Interpretation of two-by-two comparison based on 2-sided 5% significance level without correction for multiplicity
Statistical Analysis 3: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.0232, t-test, 2 sided — Interpretation of two-by-two comparison based on 2-sided 5% significance level without correction for multiplicity
Statistical Analysis 4: Comparison: Glucophage XR in Overweight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.3589, t-test, 2 sided — Interpretation of two-by-two comparison based on 2-sided 5% significance level without correction for multiplicity

2. Secondary Outcome: Mean Change From Baseline at Week 16 (95% Confidence Interval) of Fasting Plasma Glucose (FPG) - Full Analysis Set
Description: Baseline was defined as the value obtained at the screening visit. FPG was measured in millimoles/Liter (mmol/L) and obtained through local laboratories.
Time Frame: Baseline to Week 16
Population: Full Analysis Set (FAS) included enrolled participants,who took at least 1 dose of drug and had at least 1 post baseline HbA1c assessment. For this outcome measure, 1, 1, and 1 normal, overweight, obese participants, respectively, were missing and were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Groups:
- Glucophage XR in Normal Weight Participants: Normal weight defined as BMI >= 18.5 kg/m^2 and < 24 kg/m^2 ).
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 110 | 110 | 111
mmol/L | -1.979 (1.7877) [-2.317 to -1.641] | -2.171 (2.1222) [-2.572 to -1.770] | -2.141 (2.0287) [-2.522 to -1.759]
Statistical Analysis 1: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.4614, ANCOVA — Interpretation based on 2-sided 5% significance level; Change from baseline in FPG at Week 16 was dependent variable, BMI was fixed main effect, baseline FPG was covariate
Statistical Analysis 2: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants; Test type: Superiority or Other; p = 0.4696, t-test, 2 sided — Interpretation of two-by-two comparison based on 2-sided 5% significance level without correction for multiplicity
Statistical Analysis 3: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.5305, t-test, 2 sided — Interpretation of two-by-two comparison based on 2-sided 5% significance level without correction for multiplicity
Statistical Analysis 4: Comparison: Glucophage XR in Overweight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.9145, t-test, 2 sided — Interpretation of two-by-two comparison based on 2-sided 5% significance level without correction for multiplicity

3. Secondary Outcome: Mean Change From Baseline at Week 16 (95% Confidence Interval) in Fasting Total Cholesterol (TC) - Full Analysis Set
Description: For fasting total cholesterol (TC), baseline is defined as Day 1 (first day of treatment). Total cholesterol was measured in millimoles per liter (mmol/L) and obtained through local laboratories.
Time Frame: Baseline to Week 16
Population: Full Analysis Set (FAS) consisted of participants who were enrolled, took at least 1 study medication and had at least 1 post baseline HbA1c assessment. For this outcome measure, 1, 3, and 8 normal, overweight, obese participants, respectively, were missing and were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 110 | 108 | 104
mmol/L | -0.388 (0.9164) [-0.561 to -0.214] | -0.048 (0.9560) [-0.231 to 0.134] | -0.144 (0.8188) [-0.304 to 0.015]
Statistical Analysis 1: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.0305, ANCOVA — Interpretation based on 2-sided 5% significance level; Change from baseline in TC at Week 16 was dependent variable, BMI was fixed main effect, baseline TC was covariate
Statistical Analysis 2: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants; Test type: Superiority or Other; p = 0.0080, t-test, 2 sided — Interpretation of two-by-two comparison based on 2-sided 5% significance level without correction for multiplicity. For lipids, no comparison between overweight and obese was performed
Statistical Analysis 3: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.0422, t-test, 2 sided — [p-value comment as in outcome 3, analysis 2]

4. Secondary Outcome: Mean Change From Baseline at Week 16 (95% Confidence Interval) in Fasting Low-density Lipoprotein Cholesterol (LDL-C) - Full Analysis Set
Description: Baseline was defined as values obtained on Day 1. Low-density lipoprotein cholesterol (LDL-C) was measured in millimoles per liter (mmol/L) and obtained through local laboratories.
Time Frame: Baseline to Week 16
Population: Full Analysis Set (FAS) consisted of participants who were enrolled, took at least 1 study medication and had at least 1 post baseline HbA1c assessment. For this outcome measure, 1, 3, and 9 normal, overweight, obese participants, respectively, were missing and were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 110 | 108 | 103
mmol/L | -0.306 (0.5746) [-0.415 to -0.198] | -0.143 (0.6605) [-0.269 to -0.017] | -0.181 (0.6258) [-0.303 to -0.059]
Statistical Analysis 1: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.4508, ANCOVA — Interpretation based on 2-sided 5% significance level; Change from baseline in LDL-C at Week 16 was dependent variable, BMI was fixed main effect, baseline LDL-C was covariate
Statistical Analysis 2: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants; Test type: Superiority or Other; p = 0.0526, t-test, 2 sided — [p-value comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.1295, t-test, 2 sided — [p-value comment as in outcome 3, analysis 2]

5. Secondary Outcome: Mean Change From Baseline at Week 16 (95% Confidence Interval) in Fasting High-density Lipoprotein Cholesterol (HDL-C) - Full Analysis Set
Description: Baseline was defined as value obtained on Day 1 (first day of treatment). High-density lipoprotein cholesterol (HDL-C) was measured in millimoles per liter (mmol/L) and obtained through local laboratories.
Time Frame: Baseline to Week 16
Population: Full Analysis Set (FAS) consisted of participants who were enrolled, took at least 1 study medication and had at least 1 post baseline HbA1c assessment. For this outcome measure, 2, 3, and 8 normal, overweight, obese participants, respectively, were missing and were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 109 | 108 | 104
mmol/L | 0.056 (0.2016) [0.017 to 0.094] | 0.024 (0.3428) [-0.042 to 0.089] | 0.032 (0.2042) [-0.007 to 0.072]
Statistical Analysis 1: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.1431, ANCOVA — Interpretation based on 2-sided 5% significance level; Change from baseline in HDL-C at Week 16 was dependent variable, BMI was fixed main effect, baseline HDL-C was covariate
Statistical Analysis 2: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants; Test type: Superiority or Other; p = 0.4066, t-test, 2 sided — [p-value comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.4071, t-test, 2 sided — [p-value comment as in outcome 3, analysis 2]

6. Secondary Outcome: Mean Change From Baseline at Week 16 (95% Confidence Interval) in Fasting Triglycerides (TG) - Full Analysis Set
Description: Baseline was defined as value obtained on Day 1 (first day of treatment). Triglycerides (TG) were measured in millimoles per liter (mmol/L)and values obtained through local laboratories.
Time Frame: Baseline to Week 16
Population: Full Analysis Set (FAS) consisted of participants who were enrolled, took at least 1 study medication and had at least 1 post baseline HbA1c assessment. For this outcome measure, 1, 4, and 8 normal, overweight, obese participants, respectively, were missing and were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 110 | 107 | 104
mmol/L | -0.172 (2.0678) [-0.563 to 0.219] | 0.262 (3.3195) [-0.374 to 0.898] | -0.041 (2.2018) [-0.470 to 0.387]
Statistical Analysis 1: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.0210, ANCOVA — Interpretation based on 2-sided 5% significance level; Change from baseline in TG at Week 16 was dependent variable, BMI was fixed main effect, baseline TG was covariate
Statistical Analysis 2: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Overweight Participants; Test type: Superiority or Other; p = 0.2507, t-test, 2 sided — [p-value comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Glucophage XR in Normal Weight Participants vs Glucophage XR in Obese Participants; Test type: Superiority or Other; p = 0.6546, t-test, 2 sided — [p-value comment as in outcome 3, analysis 2]

7. Secondary Outcome: Mean Change From Baseline at Week 16 (95% Confidence Interval) in C-Reactive Protein (CRP) - Full Analysis Set
Description: Baseline was defined as value obtained on Day 1 (first day of treatment). C-Reactive Protein (CRP) was measured in milligrams/liter (mg/L) and values were obtained through a central laboratory; normal was less than 5.0 mg/L.
Time Frame: Baseline to Week 16
Population: Full Analysis Set (FAS) consisted of participants who were enrolled, took at least 1 study medication and had at least 1 post baseline HbA1c assessment. For this outcome measure, 102, 95, and 85 normal, overweight, obese participants, respectively, were missing and were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 9 | 16 | 27
mg/L | -0.589 (1.0914) [-1.428 to 0.250] | 3.144 (16.4019) [-5.596 to 11.884] | 1.633 (8.0706) [-1.559 to 4.826]

8. Secondary Outcome: Mean Change From Baseline at Week 16 (95% Confidence Interval) in Plasminogen Activator Inhibitor-1 (PAI-1) - Full Analysis Set
Description: Baseline was defined as value obtained on Day 1 (first day of treatment). PAI-1 (activity) was measured in units/milliliter (U/mL)and values obtained through a central laboratory; normal was less than 25.00 U/mL.
Time Frame: Baseline to Week 16
Population: Full Analysis Set (FAS) population = 111, 111, 112 in normal, overweight, obese participants respectively. For this outcome measure, 84, 79, and 75 normal, overweight, obese participants, respectively, were missing and were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 27 | 32 | 37
U/mL | 0.465 (8.5233) [-2.907 to 3.837] | 1.177 (8.9405) [-2.047 to 4.400] | -1.792 (7.9231) [-4.434 to 0.849]

9. Secondary Outcome: Mean Change From Baseline at Week 16 (95% Confidence Interval) in Adiponectin - Full Analysis Set
Description: Baseline was defined as value obtained on Day 1 (first day of treatment). Adiponectin was measured in milligrams/liter (mg/L) and values obtained through a central laboratory; normal range was 1.20 to 20.00 mg/L.
Time Frame: Baseline to Week 16
Population: Full Analysis Set (FAS) included participants who were enrolled, took at least 1 study medication and had at least 1 post baseline HbA1c assessment. For this outcome measure, 78, 70, and 72 normal, overweight, obese participants, respectively, were missing and were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 33 | 41 | 40
mg/L | 1.742 (8.6503) [-1.325 to 4.810] | 1.102 (2.2116) [0.404 to 1.801] | 0.050 (3.5516) [-1.086 to 1.186]

10. Other Pre Specified Outcome: Number of Participants With Episodes of Lactic Acidosis or Hypoglycemia From Day 1 to Week 16 - Safety Population
Description: Day 1 was first day of treatment. Lactic acidosis defined as elevated blood lactate levels (>5 mmol/L), decreased blood pH, electrolyte disturbances with an increased anion gap, and increased lactate/pyruvate ratio. Hypoglycemia (low levels of blood glucose) was reported as an adverse event. Safety population included participants who had enrolled in the study and took at least 1 dose of glucophage extended release (glucophage XR). If a subject experienced more than one adverse event, the subject was counted once at the highest severity.
Time Frame: Day 1 to Week 16
Population: All participants enrolled in the study and who received at least 1 dose of Glucophage XR.
Measure: Number; unit: participants
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 125 | 122 | 124
participants
  Lactic Acidosis | 0 | 0 | 0
  Hypoglycemia | 1 | 0 | 0

11. Other Pre Specified Outcome: Number of Participants With Clinically Significant Changes From Baseline at Week 16 in the Hematology Laboratory Test Profile - Safety Population
Description: Hematology profile = hematocrit, hemoglobin, red blood cell count (RBC), white blood cell count(WBC), lymphocytes, monocytes, basophils, eosinophils, neutrophils, platelet count. Baseline: value obtained at screening or last value obtained before treatment. LLN=lower limit of normal; ULN=upper limit of normal; preRX=pretreatment. Hemoglobin (g/dL): >3 g/dL decrease from preRX; hematocrit (%): <0.75*preRX; RBC (*10^6 c/uL): <0.75*preRX; platelet count (*10^9 c/uL): <0.67*LLN or >1.5*ULN, of if preRX<LLN, use 0.5*preRX and <100,000/mm^3; WBC (*10^3 c/uL): <0.75*LLN or >1.25*ULN, or if preRX <LLN, use <0.8*preRX or >ULN, or if preRX>ULN, use >1.2*preRX or <LLN; neutrophils+bands (*10^3 c/uL): if value <1.0*10^3 c/uL; eosinophils (*10^3 c/uL): if value >0.750*10^3 c/uL; basophils (*10^3 c/uL): if value >400/mm^3; monocytes (*10^3 c/uL): if value >2000/mm^3; lymphocytes (*10^3 c/uL): if value <0.750*10^3 c/uL or if value >7.50*10^3 c/uL.
Time Frame: Baseline to Week 16
Population: Safety population included participants who enrolled in the study and took at least 1 dose of Glucophage XR.
Measure: Number; unit: participants
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 125 | 122 | 124
participants | 0 | 0 | 0

12. Other Pre Specified Outcome: Number of Participants Who Had Abnormal Increase From Baseline at Week 16 in Kidney or Liver Function Serum Chemistry Values - Safety Population
Description: Baseline defined as value obtained either in screening visit or last value obtained before glucophage XR treatment given on Day 1. Serum chemistries evaluating kidney or liver function: blood urea nitrogen(BUN), serum creatinine (SCr), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), total bilirubin (BR), uric acid (UA). Abnormal increase in kidney and liver function tests defined as 1.25 - less than, equal to (<=)2.6 times (x) upper limit of normal (ULN)in ALT, AST, total BR, UA; abnormal increase defined as 1.25 to <= 5.1 x ULN in BUN. Safety population included participants who enrolled in the study and took at least 1 dose of Glucophage XR.
Time Frame: Baseline to Week 16
Population: Number of participants (normal, overweight, obese, respectively) who were missing values and were not included in the Week 16 analysis for the following serum chemistry tests: ALT = 14, 11, 13; AST = 14, 11, 13; total BR = 14, 11, 13; creatinine = 14, 12, 13; BUN = 14, 12, 13; UA = 14, 12, 13.
Measure: Number; unit: participants
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 125 | 122 | 124
participants
  Number with Week 16 ALT 1.25 to <= 2.6xULN | 2 | 11 | 9
  Number with Week 16 ALT > 2.6 x ULN | 0 | 0 | 0
  Number with Week 16 AST 1.25 to <= 2.6xULN | 0 | 5 | 4
  Number with Week 16 AST > 2.6 x ULN | 0 | 0 | 0
  Number with Week 16 Total BR 1.25 to <=2.6xULN | 3 | 2 | 1
  Number with Week 16 Total BR > 2.6 x ULN | 0 | 0 | 0
  Number with Week 16 BUN1.25 to <=5.1xULN | 0 | 1 | 0
  Number with Week 16 BUN > 5.1 x ULN | 0 | 0 | 0
  Number with Week 16 UA 1.25 to <=2.6xULN | 3 | 5 | 7
  Number with Week 16 UA > 2.6 x ULN | 0 | 0 | 0
  Number with Week 16 SCr 1.25 to <=2.6xULN | 0 | 0 | 0
  Number with Week 16 SCr > 1.25 x ULN | 0 | 0 | 0

13. Other Pre Specified Outcome: Number of Participants With Clinically Significant Changes From Baseline at Week 16 in Urinalysis - Safety Population
Description: Urinalysis included pH and specific gravity. Baseline defined as values obtained at screening visit. Clinically significant: outside the reference range (low/high)and judged to be significant by the investigator: Specific gravity 1.003 - 1.035; ph 5 - 8. Safety population included participants who enrolled in the study and took at least 1 dose of Glucophage XR.
Time Frame: Baseline to Week 16
Measure: Number; unit: participants
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 125 | 122 | 124
participants | 0 | 0 | 0

14. Other Pre Specified Outcome: Mean Change From Baseline at Week at Week 16 in ECG Parameter Heart Rate (HR) - Safety Population
Description: Baseline was defined as ECG obtained at the screening visit. ECG was 12-lead. Heart rate (HR) was measured in beats per minute (beats/min). Safety population included participants who enrolled in the study and took at least 1 dose of Glucophage XR.
Time Frame: Baseline to Week 16
Population: Safety population included 125, 122, 124 participants in each arm, respectively. Participants missing from analysis for change at Week 16 for Heart Rate were 17, 18, 20 participants in the normal, overweight, obese arms, respectively.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 108 | 104 | 104
beats/min | 0.4 (8.91) | 1.2 (9.56) | 1.1 (12.36)

15. Other Pre Specified Outcome: Mean Change From Baseline at Week 16 in Diastolic and Systolic Blood Pressure - Safety Population
Description: Baseline was defined as the value obtained at screening or value obtained on Day 1 before treatment. Diastolic and systolic blood pressure was measured in millimeters of mercury (mm Hg). Safety population included participants who enrolled in the study and took at least 1 dose of Glucophage XR.
Time Frame: Baseline to Week 16
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 125 | 122 | 124
mm Hg
  Week 16 change in diastolic blood pressure | -2.2 (8.63) | -4.1 (9.31) | -1.4 (9.37)
  Week 16 change in systolic blood pressure | -4.6 (14.21) | -5.5 (12.14) | -1.7 (14.55)

16. Other Pre Specified Outcome: Number of Participants Who Had a Normal Electrocardiogram (ECG) at Baseline and an ECG at Week 16 (or Termination Visit) Which Was Considered to be Abnormal With Clinical Significance - Safety Population
Description: Baseline was defined as ECG obtained at the screening visit. A judgment of clinical significance was at the discretion of the investigator. Safety population included participants who enrolled in the study and took at least 1 dose of Glucophage XR.
Time Frame: Baseline to Week 16
Population: number of participants with a normal ECG at baseline for normal weight, overweight, and obese arms were 71, 62, 65, respectively.
Measure: Number; unit: participants
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Number analyzed (Participants) | 125 | 122 | 124
participants | 0 | 1 | 3

ADVERSE EVENTS:
Time Frame: 16 Weeks
Description: A treatment-emergent AE (TEAE) was defined as an event that occurs during the treatment period.
Arm/Group | Glucophage XR in Normal Weight Participants | Glucophage XR in Overweight Participants | Glucophage XR in Obese Participants
Serious Adverse Events (participants affected / at risk) | 1/125 | 0/122 | 1/124
Other Adverse Events (participants affected / at risk) | 43/125 | 47/122 | 46/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glucophage XR in Normal Weight Participants (N=125) | Glucophage XR in Overweight Participants (N=122) | Glucophage XR in Obese Participants (N=124)
Right upper lung cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — SAE was moderate in severity and not related to treatment
Hypertension (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — SAE was moderate in severity and not considered related to treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glucophage XR in Normal Weight Participants (N=125) | Glucophage XR in Overweight Participants (N=122) | Glucophage XR in Obese Participants (N=124)
Diarrhea (Gastrointestinal disorders) | 18 (20) | 12 (17) | 4 (6)
Abdominal discomfort (Gastrointestinal disorders) | 2 (4) | 13 (14) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 6 (8) | 9 (13) | 2 (3)
Dizziness (Nervous system disorders) | 6 (9) | 4 (7) | 4 (5)
Nausea (Gastrointestinal disorders) | 2 (4) | 5 (5) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5) | 3 (3) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 6 (6)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (3)
Upper Respiratory Tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Lipid metabolism disorder (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Epigastric discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Asthenia (General disorders) | 2 (2) | 2 (3) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 3 (3) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
palpitations (Cardiac disorders) | 6 (6) | 4 (5) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
eyelid edema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
breath odor (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
feces hard (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
hypoesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
hunger (General disorders) | 1 (1) | 2 (3) | 0 (0)
thirst (General disorders) | 1 (1) | 1 (1) | 0 (0)
nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
blood lactate dehydrogenase (Investigations) | 1 (1) | 0 (0) | 0 (0)
blood uric acid increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
plasminogen activator inhibitor increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
white blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
hypoglycemia (Investigations) | 1 (3) | 0 (0) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
headache (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
toothache (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
High Density Lipoprotein cholesterol decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
hypertriglyceridemia (Investigations) | 0 (0) | 0 (0) | 2 (2)
hypocalcemia (Investigations) | 0 (0) | 0 (0) | 1 (1)
lactose intolerance (Investigations) | 0 (0) | 0 (0) | 1 (4)
musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 1 (2)
insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
rhinorrhoea (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.